CLINICAL TRIAL: NCT02520336
Title: Active Management of Postpartum Diabetes Screening After Gestational Diabetes: a Randomized Controlled Trial
Brief Title: Postpartum Diabetes Screening in Women With Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7797
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

ARMS (2):
- active management (Experimental): Laboratoy test request given postpartum with phone reminder prior to test
  Interventions: Behavioral: Reminder
- Routine care (No Intervention)

INTERVENTIONS:
Behavioral: Reminder
  Arms: active management

SUMMARY:
Assess postpartum diabetes screening in GDM patients with initiation of a reminder system in the postpartum period

ELIGIBILITY:
Inclusion Criteria: GDM, english speaking -

Exclusion Criteria: Non english speaking. Younger than 18 years of age

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Postpartum Diabetes screening in GDM patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States